CLINICAL TRIAL: NCT06666543
Title: Becoming HIV-Exposed, Uninfected Children Born to HIV-Positive Mothers Followed at Bichat Claude Bernard Hospital
Acronym: ENIVIH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231638; 2023-A02060-45 (Other: ID-RCB)
Record Dates: First submitted 2024-10-18; First posted 2024-10-30 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Virus-HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women Living with HIV: Women Living with HIV Who Have Given Birth to HIV-Exposed, Uninfected Children
  Interventions: Other: Questionary

INTERVENTIONS:
Other: Questionary — The questionnaire will address the following topics for each child who is not infected with HIV and was born to an infected mother at the time of birth:
  * Pregnancy progression
  * Immediate postpartum course
  * Medical development of the child from 0 to 3 years
  * Medical development of the child from 3 to a maximum of 15 years

SUMMARY:
"The strategies for the Prevention of Mother-to-Child Transmission of the Human Immunodeficiency Virus (HIV) are very effective and have become common practices in many contexts.

Some studies have identified clinical and biological anomalies in a small proportion of infants exposed to antiretrovirals. Beyond 2 years of age, there are few studies with low power describing the long-term consequences of perinatal exposure to antiretrovirals.

It is necessary to understand the impact of antiretroviral treatment during the perinatal period in order to improve the management of children born to HIV-positive mothers.

Retrospective cohort study with interviews of women living with HIV who were followed for a pregnancy in the Infectious diseases department of Bichat-Claude Bernard Hospital, PARIS, France.

After recruitment during a follow-up consultation:

* Information regarding the prenatal and perinatal management of HIV and the infant's outcomes up to 12 months will be collected retrospectively through the medical record
* Information regarding the child's development and follow-up from the age of 1 to a maximum of 15 years will be gathered retrospectively through a self-administered questionnaire or a questionnaire filled out with assistance during a single 1-hour interview with the mother."

DETAILED DESCRIPTION:
The latest WHO report shows that with 1.3 million (between 970,000 and 1.6 million) HIV-positive pregnant women worldwide in 2020, HIV remains a major global public health issue.

In France, about 2 per 1,000 pregnant women are infected with HIV, resulting in approximately 1,500 births per year over the past fifteen years. The administration of antiretroviral treatment to HIV-positive pregnant women and prophylaxis for infants immediately after birth is the most effective means of preventing mother-to-child transmission (MTCT) of HIV. This risk has been estimated at 0.2% during the period from 2011 to 2017 among women included in the French perinatal survey.

While the number of children infected with HIV is decreasing due to wider access to antiretroviral treatments during pregnancy, the number of HIV-exposed but uninfected children is increasing, raising questions about their long-term outcomes.

Some historical studies have identified clinical and biological anomalies, including lactic acidosis, cardiomyopathy, and neurological anomalies, suggesting mitochondrial dysfunction in a small proportion of uninfected children exposed to antiretrovirals.

Since then, recent studies have provided new evidence suggesting that HIV-exposed but uninfected children, while avoiding vertical transmission of HIV, are at a higher risk of suboptimal health outcomes, including higher rates of severe infectious morbidity, lower early childhood survival, and more frequent occurrences of growth delay and neurological development issues compared to children born without HIV exposure.

Additionally, concerns have been raised about neural tube closure anomalies in children exposed to efavirenz and dolutegravir at the time of conception. However, recent data showed that the prevalence of neural tube closure anomalies did not differ significantly between dolutegravir and other antiretrovirals since conception.

Nonetheless, some studies have acknowledged methodological weaknesses, indicating that further research is needed to evaluate each medication individually and how antiretroviral treatment regimens affect the outcomes of infants during the perinatal period.

Consensus guidelines recommend follow-up for HIV-exposed but uninfected children up to 24 months of age. Currently, there is no active long-term follow-up program in France for asymptomatic children. Follow-up may be extended if the child presents a clinical or biological anomaly. Families should be informed of the importance of reporting significant clinical events to their healthcare provider and/or the center that monitored the child in the early months of life. The healthcare provider managing the mother may also play a role in the long-term screening of significant clinical events in the child by gathering information from the mother he or she follows.

Beyond 2 years of age, there are few studies with low power describing the long-term consequences of in utero or perinatal exposure to antiretrovirals.

The participation of children and their parents in observational studies is essential for research, necessary to monitor and identify long-term health outcomes following perinatal exposure to HIV and antiretrovirals.

The objective of this retrospective study is to describe the outcomes of HIV-exposed but uninfected children born to HIV-positive mothers followed at Bichat-Claude Bernard Hospital

ELIGIBILITY:
"Inclusion Criteria

* Woman living with HIV followed for HIV infection at Bichat-Claude Bernard Hospital
* Age ≥ 18 years
* Having given birth at the maternity ward of Bichat-Claude Bernard Hospital between 01/01/2007 and 31/12/2022 to at least one child who is HIV-uninfected
* Information provided about the study and the right to refuse participation

Exclusion Criteria

* Refusal to participate in the study
* Not speaking French"

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: woman followed in the SMIT of Bichat-Claude Bernard Hospital, who gave birth at the maternity ward of this hospital between 01/01/2007 and 31/12/2022 to a child who is HIV-uninfected
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Description of clinical events of interest in children from birth until inclusion in the study (and up to a maximum age of 15 years) | 1 day
  Clinical events of interest will be collected through a survey from the mother (Eye disorders, Developmental disorders, Language disorders, Hearing disorders, Bone and joint disorders, Cardiac anomalies, Metabolic anomalies (Diabetes, Thyroid, etc.), Pulmonary anomalies, Urinary anomalies, Renal anomalies, Hematological anomalies (sickle cell disease, anemia, etc.))

SECONDARY OUTCOMES:
Describe the course of the pregnancy | at inclusion
Describe the course of the immediate postpartum period | at inclusion
Describe the medical follow-up of children between 0 and 3 years old | at inclusion
Describe the medical follow-up of children between 3 and 15 years old | at inclusion
Describe the events that occurred in children by age group | at inclusion
  events are :Eye disorders, Developmental disorders, Language disorders, Hearing disorders, Bone and joint disorders, Cardiac anomalies, Metabolic anomalies (Diabetes, Thyroid, etc.), Pulmonary anomalies, Urinary anomalies, Renal anomalies, Hematological anomalies (sickle cell disease, anemia, etc.)
Describe the events that occurred in children by type of disorders | at inclusion
  events are :Eye disorders, Developmental disorders, Language disorders, Hearing disorders, Bone and joint disorders, Cardiac anomalies, Metabolic anomalies (Diabetes, Thyroid, etc.), Pulmonary anomalies, Urinary anomalies, Renal anomalies, Hematological anomalies (sickle cell disease, anemia, etc.)
Describe the reasons for non-inclusions | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Bachelard, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France